CLINICAL TRIAL: NCT06263985
Title: Prospective Analysis of Axis(TM) Solvent-dehydrate Dermal Allograft in the Treatment of Pelvic Organ Prolapse.
Brief Title: Axis(TM) Solvent-dehydrate Dermal Allograft in the Treatment of Pelvic Organ Prolapse.
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Michigan Institution of Women's Health PC (Other)
Collaborators: Coloplast A/S (Industry)
Responsible Party: Principal Investigator, Salil Khandwala, Medical director, Michigan Institution of Women's Health PC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20214133
Record Dates: First submitted 2024-02-01; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Subjects undergoing the treatment for pelvic organ prolapse with Axis Dermis biologic mesh.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects undergoing a pelvic organ prolapse repair procedure using Axis Dermis biologic mesh (Other): This is a single are which will be composed of subjects with Stage II or greater pelvic organ prolapse who have agreed to undergoing a pelvic organ prolapse repair procedure using Axis Dermis biologic mesh. They will undergo the procedure and be followed for a period of 3 years.
  Interventions: Device: Axis Dermis biologic mesh repair for pelvic organ prolapse

INTERVENTIONS:
Device: Axis Dermis biologic mesh repair for pelvic organ prolapse — Subjects with pelvic organ prolapse will undergo a pelvic organ prolapse repair with the use of Axis Dermis biologic mesh.

SUMMARY:
The goal of this study is to assess improvement in subjects who have undergone Axis Dermis, biologic mesh for pelvic organ prolapse repair. [describe participant population/health conditions]. The main question[s] it aims to answer are:

* Is the leading edge of the prolapse above the hymen
* Does subject notice a bulge Participants will undergo Axis Dermis pelvic organ prolapse repair procedure.

DETAILED DESCRIPTION:
This is a prospective single-arm study of 50 subjects undergoing pelvic organ prolapse repair using the Axis™ Dermis biologic mesh. They will be followed for a period of 3 years. A subgroup analysis is for patients with uterine prolapse and vaginal mesh hysteropexy.

Clinical examination including vaginal wall retraction with or without pelvic ultrasound, POP-Q, and also specific validated questionnaires at baseline, 1 month, 6 month, 12 month, 24 month and 36 month visits will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with preoperative stage II or greater prolapse on the Pelvic Organ Prolapse Quantification System Assessment (POP-Q)
* Subjects who have bothersome vaginal bulge based upon symptoms.
* Subjects who undergo any type of Axis Dermis surgery (anterior, posterior, total, with or without a uterus).

Exclusion Criteria:

* Subjects who are unable to follow-up.
* Subjects who cannot complete the validated questionnaires.
* Subjects that lack competency of the English language.
* Subjects who decline to be part of the clinical trial.
* Subjects who do not sign an informed consent.

Ages: 21 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in function | Preoperative to 3 years postoperative.
  Determine improvement in function based on questionnaire Pelvic Floor Distress Inventory Q#3 "Do you usually have a bulge or something falling out that you can see or fell in the vaginal area?" Answered No, or if Yes: Not at all bothersome.
Improvement in Anatomy | Preoperative to 3 years postoperative.
  To assess improvement in anatomy with success defined as the leading edge of the prolapse is above the hymen, and no reintervention (surgery or pessary) for pelvic organ prolapse.

SECONDARY OUTCOMES:
Assess complications or untoward side effects. | intraoperative to 3 years postoperative
  Assessment of intraoperative complications (such as bleeding and injuries) and post operative complications (such as de novo incontinence, de novo dyspareunia, recurrent urinary tract infections, voiding dysfunction and effect on untreated vaginal wall).

CONTACTS AND LOCATIONS:
Overall Officials: Salil Khandwala, MD, Principal Investigator — Michigan Institution of Women's Health PC
Locations (1):
- Advanced Urogynecology of Michigan, Dearborn, Michigan, United States